CLINICAL TRIAL: NCT00088907
Title: Phase III Randomized, Placebo Controlled, Trial of Docetaxel Versus Docetaxel Plus ZD1839 (Iressa, Gefitinib) in Performance Status 2 or Previously Treated Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: Phase III Trial Of Docetaxel Versus Docetaxel Plus ZD1839 In Head And Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was unlikely that the primary endpoint would be reached based on the fifth interim analysis results.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02956; ECOG-E1302 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH); NCT00695760 (obsolete NCT alias)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2013-07

CONDITIONS: Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer
Keywords: docetaxel; gefitinib; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (docetaxel and placebo) (Active Comparator): Patients receive docetaxel intravenously (IV) over 30-60 minutes on days 1, 8, and 15 and oral placebo once daily on days 1-28.
  Interventions: Drug: docetaxel; Other: placebo
- Arm II (docetaxel and gefitinib) (Experimental): Patients receive docetaxel as in arm I and oral gefitinib once daily on days 1-28.
  ZD1839 (Iressa, gefitinib) will be given at a dose of 250 mg (one tablet) orally each day starting on day 1 and continuing for days 1 to 28 of each cycle until progression.
  In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in arm I who have disease progression may receive single-agent oral gefitinib once daily until further disease progression.
  Interventions: Drug: docetaxel; Drug: gefitinib

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm I (docetaxel and placebo)
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
  Arms: Arm II (docetaxel and gefitinib)

SUMMARY:
Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining docetaxel with gefitinib may kill more tumor cells. It is not yet known whether docetaxel is more effective with or without gefitinib in treating head and neck cancer. This randomized phase III trial is studying docetaxel and gefitinib to see how well they work compared to docetaxel alone in treating patients with metastatic or locally recurrent head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the survival of poor prognosis patients with recurrent/metastatic squamous cell carcinoma of the head and neck treated with docetaxel with or without ZD1839 (Iressa, gefitinib).

SECONDARY OBJECTIVES:

I. To determine the time to progression and response rate in poor prognosis patients with recurrent/metastatic squamous cell carcinoma of the head and neck treated with docetaxel with or without ZD1839 (Iressa, gefitinib).

II. To correlate the expression and activation status of the epidermal growth factor receptor (EGFR) signaling pathway with clinical outcome in the above patient population. The following specific biomarkers will be measured by immunohistochemistry on paraffin-embedded tumor tissue: EGFR, p-EGFR, AKT, p-AKT, Transforming growth factor (TGF)-alpha, Ki-67, extracellular-signal-regulated kinase (ERK), p-ERK, p70s6, p- p70s6 , and p27.

III. To evaluate the frequency of common polymorphisms of Cytochrome P450 3A (CYP3A) and EGFR in this study population and the impact of these polymorphisms on survival, time to progression, response rate, and toxicities.

IV. To analyze docetaxel and ZD1839 (Iressa, gefitinib) pharmacokinetics and to correlate polymorphisms with pharmacokinetic variability, response, toxicity, and other endpoints.

V. To evaluate disease-related symptoms and overall quality of life among patients receiving docetaxel only to those receiving docetaxel and ZD1839 (Iressa, gefitinib).

VI. To evaluate whether additional clinical benefit associated with ZD1839 (Iressa, gefitinib) can be detected as an improvement in patient-reported symptoms on the FACT Head and Neck Symptom Index (FHNSI)-10 and GP5.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to treatment with prior chemotherapy (pretreated vs untreated), Eastern Cooperative Oncology Group (ECOG) performance status (0 vs 1 vs 2), weight loss within the past 6 months (< 5% vs ≥ 5%), and prior cetuximab treatment (yes or no). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive docetaxel intravenously (IV) over 30-60 minutes on days 1, 8, and 15 and oral placebo once daily on days 1-28.

Arm II: Patients receive docetaxel as in arm I and oral gefitinib once daily on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in arm I who have disease progression may receive single-agent oral gefitinib once daily until further disease progression (which is called step 2 in the study).

Quality of life is assessed at baseline, on days 15 and 28 of course 1, on day 28 of all subsequent courses, and at 2-4 weeks after completion of study treatment.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 330 patients (165 per treatment arm) will be accrued for this study within 31.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck; patient must not have nasopharyngeal carcinoma of histologic types World Health Organization (WHO) 2 and 3
* Metastatic or locally recurrent carcinoma of the head and neck that is considered incurable by local therapies
* Any number of prior chemotherapy or biologic/targeted therapy regimens is allowed
* No prior systemic EGFR inhibitors, such as ZD1839 (Iressa, gefitinib)/Iressa (AstraZeneca), ABX-EBX (Abgenix), MDX-447 (Medarex/Merck), OSI-774/Tarceva (OSI pharmaceuticals), C225/Cetuximab (ImClone), PKI166 (Novartis), CI-1033 (Parke-Davis), EKB-569 (Wyeth Ayerst); treatment with paclitaxel is allowed if the patient did not progress while on paclitaxel

  * NOTE: the use of cetuximab given concurrently with radiation or chemoradiotherapy for up to 9 total weekly doses, as part of initial potentially curative therapy is allowed, if completed > 6 months prior to registration
* Patients must not receiving any other investigational agent while on the study
* Patients must have either:

  * Strata A:

    * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 (in bed 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities; up and about more than 50% of waking hours), AND no prior chemotherapy for recurrent metastatic head and neck cancer OR
  * Strata B

    * PS 0-2 AND prior chemotherapy (i.e. one or more prior chemotherapy regimens (without docetaxel)) for locally recurrent/metastatic disease or exposure to prior chemotherapy (without docetaxel) as part of primary curative therapy < 6 months prior to randomization; patients who receive chemotherapy as part of potentially curative therapy of primary disease within 6 months of randomization will be considered as having prior chemotherapy for recurrent/metastatic disease, whereas patients who received chemotherapy as part of potentially curative therapy of disease > 6 months of randomization will be considered as having no prior chemotherapy for recurrent/metastatic disease
* Patients must have fully recovered from the effects of any prior surgery, chemotherapy, or radiation therapy

  * A minimum time period of 3 weeks must elapse between the completion of radiation therapy and randomization to the study
  * A minimum period of 4 weeks must elapse between the last administration of any prior chemotherapy and randomization to the study
  * At least 2 weeks must elapse between the last administration of biologic/targeted therapy and randomization to the study
  * Patients must be > 3 weeks since major surgery, or significant traumatic injury prior to randomization
* Absolute neutrophil count (ANC) >= 1500 /mm^3
* Platelets >= 100,000 /mm^3
* Hemoglobin >= 8.0 g/dl
* Bilirubin within normal limits
* Creatinine < 2.0 or creatinine clearance of > 60 ml/min
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception while on treatment and for three months after the completion of treatment
* Patients must have measurable or non-measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST); baseline measurements and evaluations must be obtained < 4 weeks of randomization; all areas of disease should be recorded and mapped out in order to assess response and uniformity of response to therapy; disease in previously irradiated sites is considered measurable if there has been unequivocal disease progression or biopsy-proven residual carcinoma following radiation therapy; persistent disease after radiotherapy must be biopsy proven at least 8 weeks after completion of radiation therapy

  * Radiographic findings are acceptable providing that clear-cut measurements can be made
* Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 5 years post diagnosis
* Drugs that are Cytochrome P450 3A4 (CYP3A4) inhibitors should be generally avoided and if possible, discontinued, 1 week prior to initiating study drug; however, if medically necessary, they can be taken with caution after consulting with the study chair
* From patients consenting to participate in the correlative studies:

  * Tissues must be submitted as outlined in Section 10; if tissue cannot be submitted, written justification must be submitted to the ECOG Pathology Coordinating Office

Exclusion criteria:

* Prior therapy with docetaxel at any time (even if part of prior curative treatment)
* Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or serious arrhythmia requiring medication
* Hypercalcemia related to head and neck cancer
* Brain metastasis
* Current peripheral neuropathy >= grade 2 at time of randomization
* Patients have co-existing condition that would preclude full compliance with the study
* Known hypersensitivity to ZD1839 (Iressa, gefitinib) or any excipients of this product; prior history of severe hypersensitivity reaction to Docetaxel or other drugs formulated with polysorbate 80
* HIV positive patient's receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with ZD1839 (Iressa, gefitinib)
* Patients have had tumor-related hemorrhagic events in the previous three months that required as major medical intervention, such as surgery or embolization
* Patients are on therapeutic anticoagulation or have tumors that are unequivocally invading major vessels (e.g. carotid artery)
* Females are pregnant or breast feeding because chemotherapy may be harmful to the fetus or the nursing infant; also, the effects of ZD1839 (Iressa, gefitinib) on the developing human fetus are unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2004-08; Primary Completion 2009-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Result] Argiris A, Ghebremichael M, Gilbert J, Lee JW, Sachidanandam K, Kolesar JM, Burtness B, Forastiere AA. Phase III randomized, placebo-controlled trial of docetaxel with or without gefitinib in recurrent or metastatic head and neck cancer: an eastern cooperative oncology group trial. J Clin Oncol. 2013 Apr 10;31(11):1405-14. doi: 10.1200/JCO.2012.45.4272. Epub 2013 Mar 4. PMID 23460714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on August 6,2004 and terminated on November 13,2008. A total of 270 patients (136 on arm I and 134 on arm II) was enrolled to first step of the study. In July 2007, registration to step 2 (single ZD1839 therapy) was suspended because other study indicated lack of good benefit/risk profile of single agent ZD1839.
Groups:
- Arm I (Docetaxel and Placebo): Patients receive docetaxel intravenously (IV) over 30-60 minutes on days 1, 8, and 15 and oral placebo once daily on days 1-28.
  In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in arm I who have disease progression may receive single-agent oral gefitinib once daily until further disease progression.
  docetaxel: Given IV
  placebo: Given orally
- Arm II (Docetaxel and Gefitinib): Patients receive docetaxel as in arm I and oral gefitinib once daily on days 1-28.
  In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in arm I who have disease progression may receive single-agent oral gefitinib once daily until further disease progression.
  docetaxel: Given IV
  gefitinib: Given at a dose of 250 mg (one tablet) orally each day starting on day 1 and continuing for days 1 to 28 of each cycle until progression.
Period: Randomized Study (Step 1)
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib)
Started | 136 | 134
Treated | 129 | 124
Eligible | 117 | 122
Eligible and Treated | 117 | 122
Completed | 0 (Treatment would continue until disease progression, no certain fixed number of cycles.) | 0 (Treatment would continue until disease progression, no certain fixed number of cycles)
Not Completed | 136 | 134
Not completed — Lack of Efficacy | 55 | 62
Not completed — Adverse Event | 14 | 19
Not completed — Death | 11 | 12
Not completed — Withdrawal by Subject | 10 | 15
Not completed — complicating disease | 3 | 1
Not completed — unknown/not specify | 24 | 13
Not completed — ineligible or not start protocol therapy | 19 | 12
Period: Single Gefitinib Treatment (Step 2)
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib)
Started | 24 (Patients on Arm I could cross over to gefitinib after disease progression on step 1.) | 0 (Cross over to single gefitinib therapy at progression was allowed for patients on Arm I only.)
Treated | 19 | 0
Completed | 0 | 0
Not Completed | 24 | 0
Not completed — Lack of Efficacy | 16 | 0
Not completed — Death | 1 | 0
Not completed — unknown/not specify | 2 | 0
Not completed — not start protocol therapy | 5 | 0

BASELINE CHARACTERISTICS:
Population: The primary population was eligible and treated patients in the study. All study results were based on the primary population except for adverse event results. In total, 136 patients enrolled on arm I, but 19 patients were ineligible/no protocol therapy. 134 patients entered arm II, 12 of them were not eligible/not starting protocol therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib) | Total
Number analyzed (Participants) | 117 | 122 | 239
Age, Continuous [Median (Full Range); unit: years] | 61 [28 to 86] | 60 [41 to 84] | 60 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 92 | 98 | 190

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as time from registration to death from any cause. All eligible and treated patients were included in the analysis.
Time Frame: assessed every 3 months if patient is < 2 years from study entry then every 6 months if patient is 2-5 years from study entry. No specific requirements if patient is more than 5 years from study entry.
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib)
Number analyzed (Participants) | 117 | 122
months | 5.98 [4.93 to 7.43] | 7.33 [5.75 to 8.44]
Statistical Analysis 1: Comparison: Arm I (Docetaxel and Placebo) vs Arm II (Docetaxel and Gefitinib); Test type: Superiority or Other; p = 0.60, Log Rank

2. Secondary Outcome: Time to Progression
Description: Time to progression is defined as time from registration to disease progression. Disease progression was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions .
  Tumor measurements may be made using physical examination, CT scans or MRI scans. While on protocol treatment, tumor measurement by physical examination to be done every 4 weeks, and tumor measurement by CT/MRI scans to be done every 8 weeks (every 2 treatment cycles).
  All eligible and treated patients were included in the analysis.
Time Frame: as for outcome 1
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib)
Number analyzed (Participants) | 117 | 122
months | 2.14 [1.97 to 3.48] | 3.55 [2.76 to 3.75]
Statistical Analysis 1: Comparison: Arm I (Docetaxel and Placebo) vs Arm II (Docetaxel and Gefitinib); Test type: Superiority or Other; p = 0.19, Log Rank

3. Secondary Outcome: Overall Response Rate
Description: Tumor response was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Complete response (CR) was defined disappearance of all tumor lesions. Partial response (PR) was defined as as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. Overall response rate= CR+PR.
  Tumor measurements may be made using physical examination, CT scans or MRI scans. While on protocol treatment, tumor measurement by physical examination to be done every 4 weeks, and tumor measurement by CT/MRI scans to be done every 8 weeks (every 2 treatment cycles).
  All eligible and treated patients were included in the analysis.
Time Frame: as for outcome 1
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Docetaxel and Placebo) | Arm II (Docetaxel and Gefitinib)
Number analyzed (Participants) | 117 | 122
percentage of participants | 4.3 [1.4 to 9.7] | 9.8 [5.2 to 16.6]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle = 4 weeks) while on treatment and for the 30 days following the last dose of protocol drug (which was included in the form for the last cycle).
Description: Prior to diagnosis of progression / relapse or after start of non-protocol therapy, severe (Grade ≥ 3) long term toxicity that has not been previously reported was included in the report as well.
Groups:
- Step 1: Docetaxel+Placebo: * Premedication: Dexamethasone
  * Docetaxel as a 60 m inute infusion 35mg/m2 to be given on days 1,8,and 15 of a 28-day schedule
  * Placebo one tablet daily orally starting on day 1. Treatment to continue from days 1-28 of each cycle.
- Step 1: Docetaxel+ZD1839: * Premedication: Dexamethasone
  * Docetaxel as a 60 m inute infusion 35mg/m2 to be given on days 1,8, and 15 of a 28-day schedule.
  * ZD1839 (Iressa, gefitinib) 250 mg/daily orally starting on day 1. Treatment to continue from days 1-28 of each cycle.
- Step 2: ZD1839: ZD1839 (Iressa, gefitinib) 250 mg/daily orally starting on day 1. Treatment to continue from days 1-28 of each cycle.
Arm/Group | Step 1: Docetaxel+Placebo | Step 1: Docetaxel+ZD1839 | Step 2: ZD1839
Serious Adverse Events (participants affected / at risk) | 64/129 | 61/124 | 2/19
Other Adverse Events (participants affected / at risk) | 16/129 | 25/124 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Docetaxel+Placebo (N=129) | Step 1: Docetaxel+ZD1839 (N=124) | Step 2: ZD1839 (N=19)
Anaphylaxis (Immune system disorders) | 2 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 0 | 0
White blood cell decreased (Investigations) | 5 | 6 | 0
Lymphocyte count decreased (Investigations) | 9 | 4 | 0
Neutrophil count decreased (Investigations) | 4 | 4 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 3 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Fatigue (General disorders) | 21 | 14 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Weight loss (Investigations) | 2 | 1 | 0
INR increased (Investigations) | 1 | 0 | 0
Activated partial thromboplastin time pr (Investigations) | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecif (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sudden death NOS (General disorders) | 0 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 8 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 16 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 7 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Infections and infestations - Other, spe (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, spe (Infections and infestations) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 9 | 5 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 4 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0
Edema face (General disorders) | 1 | 2 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Docetaxel+Placebo (N=129) | Step 1: Docetaxel+ZD1839 (N=124) | Step 2: ZD1839 (N=19)
Anemia (Blood and lymphatic system disorders) | 10 | 16 | 0
White blood cell decreased (Investigations) | 4 | 7 | 0
Fatigue (General disorders) | 11 | 14 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 7 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 7 | 1
Nausea (Gastrointestinal disorders) | 6 | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less